CLINICAL TRIAL: NCT02160613
Title: Effect of Periodontal Surgery on Osteoprotegerin Levels in Gingival Crevicular Fluid, Saliva and Gingival Tissues.
Brief Title: Osteoprotegerin Before and After Periodontal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of periodontology, faculty of oral and dental medicine, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: OPG_OFD
Record Dates: First submitted 2014-06-07; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Periodontitis
Keywords: Osteoprotegerin; Biomarker; Chronic periodontitis; Open flap debridement
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open flap for periodontitis patients (Other): Open flap debridement
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Procedure: Open flap debridement — an access flap

SUMMARY:
The study hypothesis:

Is Osteoprotegerin a diagnostic and/or prognostic marker of periodontal disease?

DETAILED DESCRIPTION:
assessment of osteoprotegerin in patients with chronic periodontitis before and after periodontal surgery in gingival crevicular fluid, saliva and gingival tissues.

ELIGIBILITY:
Inclusion Criteria:

* severe chronic periodontitis, having pocket depth of ≥ 5 mm and clinical attachment level ≥ 5 mm

Exclusion Criteria:

* pregnant women
* subjects had <22 permanent teeth
* having any given systemic disease
* taking any type of medication and/or antibiotic therapy during the 3 months before the study
* received periodontal treatment within the past 12 months
* current or former smokers.

Ages: 32 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Osteoprotegerin levels at 3 and 6 months | Baseline, 3 months and 6 months

SECONDARY OUTCOMES:
changes from baseline in Clinical attachment level at 3 and 6 months. | Baseline, 3 months and 6 months
Changes from baseline in probing pocket depth at 3 and 6 months | baseline, 3 months and 6 months
Changes from baseline in plaque index at 3 and 6 months | baseline, 3 months and 6 months
Changes from baseline in gingival index at 3 and 6 months | baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud ElRefai, M.D., Study Director — Professor of Oral Medicine and Periodontology , Faculty of oral and dental medicine Cairo Unv.
Locations (1):
- Faculty of oral and dental medicine, Cairo, Egypt

REFERENCES:
- [Result] Liu D, Xu JK, Figliomeni L, Huang L, Pavlos NJ, Rogers M, Tan A, Price P, Zheng MH. Expression of RANKL and OPG mRNA in periodontal disease: possible involvement in bone destruction. Int J Mol Med. 2003 Jan;11(1):17-21. doi: 10.3892/ijmm.11.1.17. PMID 12469211
- [Result] Crotti T, Smith MD, Hirsch R, Soukoulis S, Weedon H, Capone M, Ahern MJ, Haynes D. Receptor activator NF kappaB ligand (RANKL) and osteoprotegerin (OPG) protein expression in periodontitis. J Periodontal Res. 2003 Aug;38(4):380-7. doi: 10.1034/j.1600-0765.2003.00615.x. PMID 12828654
- [Result] Bostanci N, Ilgenli T, Emingil G, Afacan B, Han B, Toz H, Berdeli A, Atilla G, McKay IJ, Hughes FJ, Belibasakis GN. Differential expression of receptor activator of nuclear factor-kappaB ligand and osteoprotegerin mRNA in periodontal diseases. J Periodontal Res. 2007 Aug;42(4):287-93. doi: 10.1111/j.1600-0765.2006.00946.x. PMID 17559623
- [Result] Mogi M, Otogoto J, Ota N, Togari A. Differential expression of RANKL and osteoprotegerin in gingival crevicular fluid of patients with periodontitis. J Dent Res. 2004 Feb;83(2):166-9. doi: 10.1177/154405910408300216. PMID 14742657
- [Result] Bostanci N, Ilgenli T, Emingil G, Afacan B, Han B, Toz H, Atilla G, Hughes FJ, Belibasakis GN. Gingival crevicular fluid levels of RANKL and OPG in periodontal diseases: implications of their relative ratio. J Clin Periodontol. 2007 May;34(5):370-6. doi: 10.1111/j.1600-051X.2007.01061.x. Epub 2007 Mar 13. PMID 17355365
- [Result] Buduneli N, Buduneli E, Kutukculer N. Interleukin-17, RANKL, and osteoprotegerin levels in gingival crevicular fluid from smoking and non-smoking patients with chronic periodontitis during initial periodontal treatment. J Periodontol. 2009 Aug;80(8):1274-80. doi: 10.1902/jop.2009.090106. PMID 19656027
- [Result] Costa PP, Trevisan GL, Macedo GO, Palioto DB, Souza SL, Grisi MF, Novaes AB Jr, Taba M Jr. Salivary interleukin-6, matrix metalloproteinase-8, and osteoprotegerin in patients with periodontitis and diabetes. J Periodontol. 2010 Mar;81(3):384-91. doi: 10.1902/jop.2009.090510. PMID 20192865
- [Result] Bostanci N, Saygan B, Emingil G, Atilla G, Belibasakis GN. Effect of periodontal treatment on receptor activator of NF-kappaB ligand and osteoprotegerin levels and relative ratio in gingival crevicular fluid. J Clin Periodontol. 2011 May;38(5):428-33. doi: 10.1111/j.1600-051X.2011.01701.x. Epub 2011 Jan 24. PMID 21261673
- [Result] Dereka XE, Markopoulou CE, Fanourakis G, Tseleni-Balafouta S, Vrotsos IA. RANKL and OPG mRNA level after non-surgical periodontal treatment. Inflammation. 2010 Jun;33(3):200-6. doi: 10.1007/s10753-009-9174-7. PMID 20033478
- [Derived] Hassan SH, El-Refai MI, Ghallab NA, Kasem RF, Shaker OG. Effect of periodontal surgery on osteoprotegerin levels in gingival crevicular fluid, saliva, and gingival tissues of chronic periodontitis patients. Dis Markers. 2015;2015:341259. doi: 10.1155/2015/341259. Epub 2015 Feb 28. PMID 25814780